CLINICAL TRIAL: NCT06168383
Title: A Multicenter, Double-blind, Placebo Randomized , Phase2b Study to Evaluate the Efficacy and Safety of HSK31679 in Chinese Patients With Non-Alcoholic Steatohepatitis (NASH).
Brief Title: To Evaluate the Efficacy and Safety of HSK31679 in Chinese Patients With Non-Alcoholic Steatohepatitis (NASH) .
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK31679-202
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Non-Alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Double-blind 80 mg Daily (Experimental): Patients take double-blind HSK31679 80 mg for 52 weeks
  Interventions: Drug: HSK31679 80mg
- Double-blind 160 mg Daily (Experimental): Patients take double-blind HSK31679 160 mg for 52 weeks
  Interventions: Drug: HSK31679 160mg
- Placebo (Placebo Comparator): Patients take double-blind placebo for 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK31679 80mg — once daily, oral administration of HSK31679 80mg from Day 1 to Week 52.
  Arms: Double-blind 80 mg Daily
Drug: HSK31679 160mg — once daily, oral administration of HSK31679 160mg from Day 1 to Week 52.
  Arms: Double-blind 160 mg Daily
Drug: Placebo — once daily, oral administration of placebo from Day 1 to Week 52.
  Arms: Placebo

SUMMARY:
A double-blind placebo controlled, randomized, Phase 2b study to evaluate the efficacy and safety of once-daily, oral administration of 80 or 160 mg HSK31679 versus matching placebo in Patients With Non-Alcoholic Steatohepatitis (NASH) and Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Must be willing to participate in the study and provide written informed consent.
2. Male or female aged 18 ≤ age < 65 at the time of signing the informed consent
3. Must have had prior liver biopsy within 180 days of randomization with fibrosis stage 2 to 3 and a NAS of ≥4 with at least a score of 1 in each of the lobular inflammation and ballooning degeneration.
4. Must have confirmation of ≥8% liver fat content on MRI-PDFF.
5. Weight changes≤5% in the 6 weeks prior to randomization.If a historical biopsy is to be used, patients must have had weight changed≤5%, too.

Exclusion Criteria:

1. History or presence of cirrhosis，hepatic decompensation or impairment defined as presence of any of the following: history of esophageal varices, ascites, or hepatic encephalopathy, or hepatocellular carcinoma.
2. Use of high dose vitamin E (>400 IU/day)，polyunsaturated fatty acid or ursodeoxycholic acid unless stable for ≥6 months prior to an eligible screening liver biopsy. Use of thiazolidinediones, sodium-glucose co-transporter 2 inhibitors or a complex oral anti-diabetic (OAD) regimen (3 or more OADs) unless stable for ≥3 months prior to an eligible screening liver biopsy.
3. Use of Glucagon-like peptide 1 [GLP-1] agonist therapy (e.g.,liraglutide, semaglutide, dulaglutide and exenatide ) within 6 months prior to an eligible screening liver biopsy.
4. Use of drugs that have the potential to affect thyroid hormone production and/or interfere with thyroid function.
5. Potent inhibitors of CYP2C8 such as gemfibrozil and trimethoprim are prohibited. An inducer of CYP2C8, rifampicin, is prohibited.
6. Use of drugs historically associated with NAFLD/NASH for 2 weeks prior to an eligible screening liver biopsy, which include, but are not limited, to the following: total parenteral nutritionamiodarone, methotrexate, systemic glucocorticoids (if use within 3 months prior to a biopsy is also not permitted), tamoxifen, tetracycline, estrogens at doses greater than those used for hormone replacement or contraception, anabolic steroids , valproic acid, and known hepatotoxins.
7. Regular use of drugs historically associated with NAFLD/NASH within 12 months prior to liver biopsy (including historical biopsy), which include, but are not limited, to the following:PPAR agonists (e.g. lanifibranor, Siglitazone sodium) ，FXR agonists (e.g., obecholic acid, HTD1801)，FGF21 analogs (e.g., AP025, efruxifermin , pegozafermin(B1089-1001)) ; DGAT2 inhibitors (e.g., PF 6865571 and ION224),PDE inhibitors (e.g., ZSP1601) and other thyroid hormone receptor B agonists [e.g.,resmetirom（MGL-3196）、ASC41 and VK2809).
8. Lipid-lowering therapy that did not meet the following criteria: fenofibrate, ezetimibe stable for at least 3 months before randomization and remained unchanged during study treatment, and statins stable for at least 4 weeks before randomization and remained unchanged during study treatment.
9. Type 1 diabetes or uncontrolled Type 2 diabetes defined as:

   * Hemoglobin A1c >9.5% at screening (patients with HbA1c >9.5% may be rescreened),
   * Insulin dose adjustment >20% within 60 days prior to enrollment,
   * Requirement for glucagon-like peptide analogue (unless on a stable dose ≥ 6 months prior to screening) or History of severe hypoglycemia (symptomatic hypoglycemia requiring outside assistance to regain normal neurologic status).
10. Uncontrolled hypertension (either treated or untreated) defined as systolic blood pressure >160 mmHg or a diastolic blood pressure >100 mmHg at screening.
11. Evidence of other forms of chronic liver disease including the following:biliary bypass, drug induced liver disease, alcoholic liver disease, autoimmune hepatitis, primary biliary cholangitis (PBC), primary sclerosing cholangitis (PSC), hemohemosis, Wilson's disease, α-1 antitrypsin deficiency, bile duct obstruction, primary or metastatic liver cancer, hepatitis B, or present Hepatitis virus (HCV) infection.
12. Thyroid diseases: hyperthyroidism and hypothyroidism. Thyroid peroxidase antibodies (TPOAb) or thyroglobulin antibodies (TGAb) that have been determined by the investigators to be clinically significant.
13. Myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass graft, or stroke within 6 months prior to screening.
14. New York Heart Association class III or IV heart failure, or known left ventricular ejection fraction <30%.
15. Serum ALT or AST >5 × ULN; Serum ALP≥2× ULN；eGFR<60 mL/min/1.73m2；INR>1.5× ULN；platelets < 80×109/L.
16. Participation in an investigational new drug trial in the 90 days prior to randomization.
17. Any other condition which, in the opinion of the Investigator, would impede compliance, hinder completion of the study, compromise the well-being of the patient, or interfere with the study outcomes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Proportions of patients(HSK31679-treated versus placebo-treated) with NASH improvement and with no worsening of fibrosis at week 52 compared with Baseline. | from Baseline to 52 weeks
  Improvement of NASH is defined as a 2-point reduction in NAS with at least 1-point reduction in ballooning and no increase in steatosis.

SECONDARY OUTCOMES:
Proportions of patients(HSK31679-treated versus placebo-treated) with improvement in liver fibrosis greater than or equal to one stage and no worsening of NASH at week 52 compared with Baseline. | from Baseline to 52 weeks
Proportions of patients(HSK31679-treated versus placebo-treated) with both improvement of NASH and fibrosis at week 52 compared with Baseline. | from Baseline to 52 weeks
The percent relative change from baseline in hepatic fat fraction by MRI-PDFF at 12, 24, 36 and 52 weeks for HSK31679 versus placebo. | from Baseline to 12, 24, 36, and 52 weeks
The proportions of patients with 30% or more relative hepatic fat reduction at 12 , 24 , 36 and 52 weeks for HSK31679 versus placebo. | from Baseline to 12, 24, 36, and 52 weeks
Assess the effect of HSK31679 compared to placebo on Parameters of blood lipids measured by percent change from Baseline to 12, 24, 36, and 52 weeks. | from Baseline to 12, 24, 36, and 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, Tsinghua University, Beijing, China